CLINICAL TRIAL: NCT03260907
Title: Efficacy and Safety of Electroacupuncture and Acupuncture in Postmenopausal Women With Overactive Bladder ; A Multicenter, Randomized, Controlled, Parallel Clinical Trial
Brief Title: Efficacy and Safety of Electroacupuncture and Acupuncture in Postmenopausal Women With Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: DongGuk University (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Jung Seunghyun, Principal Investigator, DongGuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-0008
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Overactive Bladder; Menopause
Keywords: Overactive bladder; menopause; Postmenopausal overactive bladder; Electroacupuncture
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Electroacupuncture; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture (Experimental): The patients in this group received electroacupuncture using the same acupuncture points prescribed by a certified Korean Medicine Doctor with more than 6 years of oriental medicine college education and 1 years of clinical experience.
  Interventions: Procedure: Electroacupuncture
- Acupuncture (Experimental): The patients in this group received acupuncture without electric stimulation using the same acupuncture points prescribed by a certified Korean Medicine Doctor with more than 6 years of oriental medicine college education and 1 years of clinical experience.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — The treatment is to be applied twice a week for acupuncture points(unilaterally at CV3, CV4, GV20 and bilaterally at KI3, SP6), used for all the patients assigned to this group. Disposable, sterilized, filiform acupuncture needles manufactured is to be used. An electric acupuncture device (CellMac STN-110, Stratek Co, Republic of Korea) will be connected to the CV3-CV4, KI3-SP6 acupoints and deliver stimulation with a 2-Hz frequency, asymmetric bimodal pulse, continuous wave mode, maximum intensity below the threshold (7.6~13.9mA).
  Other Names: EA
  Arms: Electroacupuncture
Procedure: Acupuncture — The treatment is to be applied twice a week for acupuncture points(unilaterally at CV3, CV4, GV20 and bilaterally at KI3, SP6), used for all the patients assigned to this group. Disposable, sterilized, filiform acupuncture needles manufactured is to be used.
  Other Names: AC
  Arms: Acupuncture

SUMMARY:
The purpose of this study is to verify the efficacy and safety of electroacupuncture treatment of postmenopausal women with overactive bladder (OAB).

DETAILED DESCRIPTION:
The investigators targeted the patients of menopausal women with OAB. After treatment in 2 groups - electroacupuncture treatment and acupuncture treatment - the investigators will compare the improvement of the urinary symptoms and the quality of life, and further the best treatment method. In addition, the investigators are going to evaluate the safety of abnormal reaction during the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women over 40 years of age without the possibility of pregnancy
2. Have a history of amenorrhea for at least 1 year and have no previous history of hormone replacement therapy for the last 6 months
3. With symptoms of urinary frequency and urgency lasting more than three months
4. Who fit the diagnostic criteria for OAB, with a total score more than three points in Korean version overactive bladder symptom score (OABSS)
5. Who have average urinary frequency of more than eight times per day and urgency which is defined as urgency rating scale (URS) on bladder diary is more than two points and/or UUI on 3-day bladder diary during one week screening period
6. Who agree to this clinical study after sufficient explanation

Exclusion Criteria:

1. Diag¬nosed with UTI by urine examination
2. With stress urinary incontinence without symptoms of OAB
3. With suspected of having voiding dys¬function induced by neurological damage
4. With a medical history of cystocele, uterine pro¬lapse or similar
5. With a medical history of obstructive uropathy such as urinary stones and urinary tumors
6. With a surgical history of urethra or bladder
7. With a medical history of malignant tumors of urinary tract
8. With a medical history of neurologic disease or psychi¬atric illness
9. Have an artificial cardiac pacemaker or implantable cardioverter defibrillator in the chest
10. Have experienced a hypersensitivity reaction after an acupuncture treatment, or show any other contraindications;
11. Who participated in another clinical trial within the past three months
12. Who have taken therapeutic drugs that may affect blad¬der function within one month of the start of this study
13. With inadequate literacy to complete study documents

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2018-03-02 (Estimated); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
3-day bladder diary change | at baseline, after 6 weeks of treatment (the end of the treatment period), after 10 weeks of treatment(follow up evaluation)
  The daytime micturitions per 24 hr, nocturnal micturitions per 24 hr, total count of urgency (sum of urgency epi¬sodes defined as URS ≥ 3 for three days), total urgency score (sum of urgency score for three days), and total count of UUI (sum of UUI episodes for three days) is checked.

SECONDARY OUTCOMES:
The overactive bladder symptom score (OABSS) change | at baseline, after 6 weeks of treatment (the end of the treatment period), after 10 weeks of treatment(follow up evaluation)
  The OABSS consists of four questions regarding OAB symptoms; day¬time frequency, nocturia, urgency, and UUI. The sum of the four scores runs between 0 and 15.
The King's Health Questionnaire (KHQ) | at baseline, after 6 weeks of treatment (the end of the treatment period), after 10 weeks of treatment(follow up evaluation)
  The KHQ is a urine questionnaire that can assess the severity of urination symptoms and evaluate the impact of urination symptoms on quality of life. This questionnaire is known to have reliability and validity in measuring the quality of life of patients with incontinence. The 10 domains from the KHQ evaluated are general health perception, incontinence impact, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep/energy, severity measures, and symptom severity.
Adverse events (AEs) | at baseline, every treatment(12 sessions in 6 weeks, including after 6 weeks of treatment (the end of the treatment period), after 10 weeks of treatment(follow up evaluation)
  Adverse events (AEs) indicate undesirable and unintentional signs, symptoms, or diseases that develop after intervention during the period of a clinical trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguk university Bundang Oriental Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nam EY, Park JY, Jo J, Jung SH, Lim CY, Kim DI. Electroacupuncture to treat with Overactive Bladder in Postmenopausal Women: study protocol for a multicenter, randomized, controlled, parallel clinical trial. Trials. 2018 Sep 15;19(1):493. doi: 10.1186/s13063-018-2715-3. PMID 30219086